CLINICAL TRIAL: NCT07295704
Title: Comparative Evaluation of Micropulse Laser in Treatment of Initial and Refractory Cases of Center-Involved Diabetic Macular Edema
Brief Title: Micropulse Laser in Treatment of Initial and Refractory Cases of Center-Involved Diabetic Macular Edema
Status: Recruiting | Type: Observational
Sponsor: The General Authority for Teaching Hospitals and Institutes (Network)
Responsible Party: Principal Investigator, Hossam Abdelfattah Husein Hassan, Fellow of Ophthalmology, Sohag Teaching Hospital, Egypt., The General Authority for Teaching Hospitals and Institutes
Other Study IDs: HSO00011
Record Dates: First submitted 2025-12-06; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Micropulse Laser; Treatment; Initial; Refractory; Center-Involved Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Naïve center-involved diabetic macular edema group: Patients with treatment-naïve center-involved diabetic macular edema.
  Interventions: Other: Micropulse Laser
- Refractory center-involved diabetic macular edema group: Patients with refractory center-involved diabetic macular edema.
  Interventions: Other: Micropulse Laser

INTERVENTIONS:
Other: Micropulse Laser — All laser procedures will be performed in a darkened room. The laser will be delivered together in an 8×8 pattern mode with high density (0µm of spacing) over the entire area of macular edema, including the foveal center and unthickened (200µm) retina with no attempt to target or avoid microaneurysms.

SUMMARY:
This study aims to evaluate the effect of subthreshold 577 nm micropulse laser photocoagulation in the treatment of initial and refractory cases of Center-Involved Diabetic Macular Edema.

DETAILED DESCRIPTION:
Diabetic Retinopathy (DR) is a common and specific microvascular complication of diabetes that affects 17-54% of people with diabetes aged between 49 and 60 years.

Diabetic macular edema (DME) is one of the most common causes of visual loss in today's society. It affects about 10% of diabetic individuals and 29% of those who have had the condition for more than 20 years.

In micropulse mode, the laser emits short pulses, thereby reducing thermal energy in the target area.

This strategy has two properties: a shorter exposure time and a subvisible clinical endpoint, delivering energy by dividing the beam into a series of short pulses (100-300 µs). Every single pulse has an "on and off" duration (duty cycle (DC)), enabling tissues to cool down before the next pulse.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Both sexes.
* Patients with type 1 or 2 diabetes mellitus (DM), best-corrected visual acuity (BCVA) of 20/400 or better, and center-involved DME [defined as a central macular thickness (CMT) of >250 but <700µm measured by spectral-domain optical coherence tomography].
* Patients with any level of non-proliferative diabetic retinopathy or proliferative diabetic retinopathy with adequate panretinal photocoagulation (PRP) and no signs of disease activity determined by fluorescein angiography (FA).

Exclusion Criteria:

* Monocular eyes.
* Chronic renal failure or renal transplant because of diabetic nephropathy.
* Glycated hemoglobin (HbA1c) of more than 10%.
* Vitreomacular traction syndrome.
* Epiretinal membrane.
* PRP within 4months before the treatment.
* Intraocular surgery within 6months, including cataract or vitreoretinal operation.
* Rubeosis iridis.
* Severe glaucoma.
* High-risk proliferative diabetic retinopathy.
* Poor dilation.
* Increased foveal avascular zone.
* Any condition that could interfere with optical coherence tomography (OCT) measurement or visual acuity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort comparative study was conducted at the Ophthalmology Department of Sohag Teaching Hospital, with approval from the institutional ethical committee.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change of best-corrected visual acuity | 6 months post-procedure
  Change of best-corrected visual acuity will be recorded.

SECONDARY OUTCOMES:
Change of central macular thickness | 6 months post-procedure
  Change of central macular thickness will be recorded.
Change of area thickness | 6 months post-procedure
  Change of area thickness will be recorded.
Change of macular volume | 6 months post-procedure
  Change of macular volume will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- the General Authority for Teaching Hospitals and Institutes, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.